CLINICAL TRIAL: NCT00991302
Title: Durability of Adherence in Self-Management of HIV
Acronym: DASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5250; 1U01AI068636 (NIH); 10654
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Results first posted 2015-08-26 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-02

CONDITIONS: HIV Infections
Keywords: Adherence; Behavioral Intervention; Antiretroviral Therapy; ART; Highly Active Antiretroviral Therapy; HAART; Treatment experienced
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CAP-IT (Experimental): Participants received the modified CAP-IT adherence intervention in addition to standard care.
  Modified client adherence profiling and intervention tailoring (CAP-IT): Interventions designed to improve medication adherence, modified to specifically target people first starting highly active antiretroviral therapy (HAART)
  Interventions: Behavioral: CAP-IT
- Standard care (No Intervention): Participants received standard care.

INTERVENTIONS:
Behavioral: CAP-IT — Interventions designed to improve medication adherence, modified to specifically target people first starting highly active antiretroviral therapy (HAART)
  Other Names: Client adherence profiling and intervention tailoring
  Arms: CAP-IT

SUMMARY:
Adherence to highly active antiretroviral therapy (HAART) is critical to successful treatment of HIV. This study tested an intervention that helps people infected with HIV take all their medications when and how they were supposed to.

DETAILED DESCRIPTION:
People infected with HIV must take the regimen of highly active antiretroviral therapy (HAART) medications as prescribed to them, without missing doses, or they risk developing a resistant strain of the virus. Resistant strains of the virus do not respond to certain HAART regimens and are more dangerous for patients. Poor HAART adherence can lead to further HIV progression, more hospitalizations and opportunistic infections, and required use of second-line therapies. Interventions to increase adherence have had mixed success, with little data to support long-term effects and no one strategy emerging that provides consistent positive effects. The client adherence profiling and intervention tailoring (CAP-IT) program was first developed to increase adherence among people already on HAART with in-home nursing. This study modified CAP-IT to treat people newly on HAART and then tested whether this modified CAP-IT improved long-term HAART adherence.

This study included two stages. The first stage consisted of two focus groups, one made up of HIV care providers and professionals and the other made up of people infected with HIV who had started HAART within the last year. Each focus group met once, for approximately 2 hours, to determine what modifications would best adapt the CAP-IT program to HIV-infected people first starting HAART.

The second stage consisted of a randomized trial comparing the modified CAP-IT program to standard of care. Participation in this stage lasted for 72 weeks. Participants were randomly assigned to receive either standard care or the modified CAP-IT program in addition to standard care. The CAP-IT program involved two steps. The first was an assessment of factors relating to adherence, and the second was development of an individualized plan to address the deficits found.

Study visits were completed at entry, at Weeks 4 and 12, and then every 12 weeks for approximately 72 weeks. Assessments for the study included a questionnaire about health attitudes, a physical exam, counting of pills, and answering questions about taking medications.

ELIGIBILITY:
Inclusion Criteria:

* Stage 1

  * HIV infected Individuals on Highly Active Antiretroviral Therapy (HAART):

    * HIV-1 infection
    * Initiated HAART within 1 year prior to study entry and remained on HAART for at least 30 consecutive days
    * Men and women who hade reached the legal age of majority in the country where they are being enrolled
    * Ability and willingness to provide informed consent
    * Willingness to discuss personal topics during an audio-taped group interview
    * Willingness to protect the confidentiality of other focus group participants
  * Health Care Providers and Professionals:

    * Healthcare providers or professionals (e.g., medical doctors [MDs], nurse practitioner [NPs], physician assistants [PAs], adherence counselors) recruited from outside of the local clinical research site (CRS) whose patient population included a majority of HIV-1 seropositive patients and who had recent experience managing ART-naive individuals starting HAART
    * Men and women who had reached the legal age of majority in the country where they are being enrolled
    * Willingness to discuss personal topics during an audio-taped group interview
    * Willingness to protect the confidentiality of other focus group participants and of the proceedings
* Stage 2:

  * HIV-1 infection
  * Antiretroviral (ARV) treatment naive, but planning to initiate HAART within 7 days of study entry either in the context of an approved parent AIDS Clinical Trial Group (ACTG) clinical trial or in the context of primary HIV care at a University of California, San Diego (UCSD), USA or Asociacion Civil Impacta Salud Y Educaci (IMPACTA), Peru, CRS-affiliated site
  * HIV-1 RNA greater than 1,000 copies/mL obtained within 90 days prior to study entry by any laboratory that has a clinical laboratory improvement amendments (CLIA) certification or its equivalent
  * CD4+/CD8+ count obtained within 90 days prior to study entry by any laboratory that has a CLIA certification or its equivalent
  * Men and women who had reached the legal age of majority in the country where they are being enrolled
  * Ability to follow instructions and complete surveys and questionnaires with minimal assistance

Exclusion Criteria:

* Stage 1

  * HIV-1 Infected Individuals on HAART:

    * Failure to remain on HAART for at least 30 consecutive days
    * Diminished cognitive capacity that, in the opinion of the screening CRS clinician, would interfere with study participation
    * Participation in any prior focus group for study A5250
  * Health Care Providers and Professionals:

    * Health care providers and professionals who would be involved in administering standard of care (SOC) treatment and adherence counseling to Stage 2 participants randomized to the SOC arm or CRS investigators or health care providers and professionals directly involved in measuring adherence outcomes in Stage 2
    * Participation in any prior focus group for study A5250
* Stage 2:

  * Potential participants who were, in the judgment of the research team, unable to complete the protocol
  * Potential participants who were starting a NNRTI-based regimen within 12 months after receiving single-dose NVP during pregnancy to prevent MTCT of HIV
  * Potential participants who were partners or close contacts of participants enrolled in Stage 2
  * Potential participants who were currently enrolled in an ACTG protocol utilizing or testing an adherence intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2010-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Constance Benson, MD, Study Chair — University of California, San Diego; Tari Gilbert, MSN, Study Chair — University of California, San Diego
Locations (2):
- Ucsd, Avrc Crs, San Diego, California, United States
- Barranco CRS (11301), Lima, Peru

REFERENCES:
- [Background] Lu M, Safren SA, Skolnik PR, Rogers WH, Coady W, Hardy H, Wilson IB. Optimal recall period and response task for self-reported HIV medication adherence. AIDS Behav. 2008 Jan;12(1):86-94. doi: 10.1007/s10461-007-9261-4. Epub 2007 Jun 19. PMID 17577653
- [Background] Wagner GJ, Kanouse DE, Golinelli D, Miller LG, Daar ES, Witt MD, Diamond C, Tilles JG, Kemper CA, Larsen R, Goicoechea M, Haubrich RH. Cognitive-behavioral intervention to enhance adherence to antiretroviral therapy: a randomized controlled trial (CCTG 578). AIDS. 2006 Jun 12;20(9):1295-302. doi: 10.1097/01.aids.0000232238.28415.d2. PMID 16816559

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CAP-IT | Standard Care
Started | 86 | 86
Completed | 72 | 73
Not Completed | 14 | 13
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 14 | 12

BASELINE CHARACTERISTICS:
Population: Intention to treat: All eligible participants were included in the baseline characteristics.
Groups:
- Total: Total of all reporting groups
Arm/Group | CAP-IT | Standard Care | Total
Number analyzed (Participants) | 86 | 86 | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (8) | 32 (10) | 31 (9)
Age, Customized [Number; unit: participants]
  18-29 years | 48 | 43 | 91
  30-39 years | 25 | 23 | 48
  40-49 years | 10 | 14 | 24
  50+ years | 3 | 6 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 6
  Male | 85 | 81 | 166
Race/Ethnicity, Customized [Number; unit: participants]
  White Non-Hispanic | 7 | 16 | 23
  Black Non-Hispanic | 4 | 1 | 5
  Hispanic (Regardless of Race) | 73 | 62 | 135
  Asian, Pacific Islander | 0 | 3 | 3
  More than Once Race | 1 | 1 | 2
  Missing | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 26 | 26 | 52
  Peru | 60 | 60 | 120
Regimen complexity [Number; unit: participants]
  QD | 25 | 25 | 50
  BID or TID | 61 | 61 | 122
HIV-1 RNA [Mean (Standard Deviation); unit: log10 copies/mL] | 4.9 (0.8) | 5.0 (0.7) | 5.0 (0.7)
CD4+ T-cell count [Mean (Standard Deviation); unit: cells/mm^3] | 318 (178) | 313 (213) | 315 (195)

OUTCOME MEASURES:

1. Primary Outcome: Mean Self-reported Adherence Score (%) Over a One-month Recall
Description: The adherence self-report questionnaire captured adherence at an Antiretroviral Therapy (ART) regimen over a one-month recall (0-100): 0 means none of anti-HIV medications were taken, 100 means every single dose of anti-HIV medications were taken. The primary endpoint evaluated for each participant was the average self-reported adherence over a one-month recall across each of their study visit week 4, 12, 24, 36, and 48: missing values were ignored.
  Note: This was a change to the primary endpoint as described in the study protocol. This was due to an update to ACTG Case Report Form (CRF) that captured self-report adherence. Since the data captured on this form captured adherence over a longer timeframe and allowed for more variability in response, it was anticipated this endpoint would provide greater power to assess treatment differences.
Time Frame: At weeks 4, 12, 24, 36, and 48
Population: Intention to treat: All eligible participants were included in the analysis: participants were analyzed per original assigned randomized treatment. Missing data were assumed missing completely at random.
Measure: Median (Inter-Quartile Range); unit: percentage of adherence score
Arm/Group | CAP-IT | Standard Care
Number analyzed (Participants) | 86 | 86
percentage of adherence score | 97.5 [93.4 to 100.0] | 98.2 [94.0 to 99.8]
Statistical Analysis 1: Comparison: CAP-IT vs Standard Care; Treatment comparison was made using a Wilcoxon rank sum test stratified by dosing complexity. The test was not stratified by region of enrollment due to dosing complexity and region of enrollment were almost identical: almost all (exception with two) participants in the US region were on QD and all participants in the Peru region were on BID or TID; Test type: Superiority or Other; p = 0.52, Wilcoxon (Mann-Whitney); stratified by dosing complexity

2. Secondary Outcome: Mean Self-reported Adherence Score Over a One-month Recall
Description: The mean of participant's average self-reported adherence score over a one-month recall across visit week 4, 12, 24, 36, 48, 60, and 72; missing values were ignored.
Time Frame: Weeks 4, 12, 24, 36, 48, 60, and 72
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of adherence score
Arm/Group | CAP-IT | Standard Care
Number analyzed (Participants) | 86 | 86
percentage of adherence score | 97.2 [92.9 to 99.4] | 97.8 [93.4 to 99.7]

3. Secondary Outcome: Kaplan-Meier Estimate of the Cumulative Probability of Time to Change of Initial Antiretroviral (ARV) Treatment Regimen for Any Reason by Week 48
Description: The Kaplan-Meier estimate of the cumulative probability of initial antiretroviral (ARV) treatment regimen for any reason by week 48.
  Time to ARV treatment regimen change was defined as first time to change in the drug class of participant's ART regimen for any reason from study entry. Participants completing the study without a change in the drug class of their ART regimen were censored at their last visit.
Time Frame: From study entry to week 48
Population: Intention to treat: All eligible participants were included in the analysis: participants were analyzed per original assigned randomized treatment.
Measure: Number (95% Confidence Interval); unit: cumulative probability per 100 persons
Arm/Group | CAP-IT | Standard Care
Number analyzed (Participants) | 86 | 86
cumulative probability per 100 persons | 17 [9 to 25] | 19 [11 to 28]

4. Secondary Outcome: Virologic Suppression
Description: Virologic suppression was defined as HIV-1 RNA <=200 copies/mL at week 24, 48, and 72. The results obtained within +/- 12 weeks of 24, 48, and 72 weeks were included. If there were multiple HIV-1 RNA measurement within the specified window, the HIV-1 RNA result closest to the center of the window was selected.
Time Frame: At week 24, 48, 72
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CAP-IT | Standard Care
Number analyzed (Participants) | 86 | 86
percentage of participants
  Week 24 (nCAP-IT=80, nSOC=79) | 94 [88 to 99] | 86 [78 to 94]
  Week 48 (nCAP-IT=77, nSOC=73) | 95 [90 to 100] | 85 [77 to 93]
  Week 72 (nCAP-IT=64, nSOC=66) | 88 [79 to 96] | 88 [80 to 96]

5. Secondary Outcome: Self-management Skills, as Measured by Self-reported General Self-efficacy Scale (GSES) Score
Description: The GSES is a 10-item scale designed to assess optimistic self-beliefs used to cope with a variety of demands in life. The scale was designed to assess self efficacy, i.e., the belief that one's actions are responsible for successful outcomes. The scaled score for each question ranges from 1 to 4. Higher scores indicate participant's stronger belief in self-efficacy.
  The GSES score was sum of all responses. The range was from 0 to 40 scores: any unfinished question got a score of zero.
Time Frame: At weeks 0 (entry), 4, 12, 24, 36, 48, 60, and 72
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | CAP-IT | Standard Care
Number analyzed (Participants) | 86 | 86
scores on a scale
  Week 0 (nCAP-IT=86, nSOC=86) | 36 [31 to 39] | 36 [32 to 38]
  Week 4 (nCAP-IT=84, nSOC=86) | 37 [33 to 38] | 36 [31 to 39]
  Week 12 (nCAP-IT=81, nSOC=77) | 36 [33 to 38] | 36 [32 to 39]
  Week 24 (nCAP-IT=81, nSOC=82) | 36 [32 to 39] | 37 [34 to 39]
  Week 36 (nCAP-IT=81, nSOC=79) | 37 [33 to 39] | 37 [33 to 39]
  Week 48 (nCAP-IT=75, nSOC=77) | 37 [34 to 40] | 38 [33 to 40]
  Week 60 (nCAP-IT=73, nSOC=73) | 37 [34 to 39] | 36 [33 to 39]
  Week 72 (nCAP-IT=71, nSOC=72) | 37 [31 to 40] | 38 [33 to 40]

6. Secondary Outcome: Cumulative Probability of First Grade 3 or 4 Adverse Events (AEs)
Description: The Kaplan-Meier estimate of the cumulative probability of experiencing a grade 3 or 4 adverse event by week 72.
  New Grade 3 or 4 signs, symptoms were identified by MedDRA preferred term. Events were included regardless of participant status on ART. If a participant had multiple reports of the same event, only the event reported at the highest grade were included.
  Time was measured from the study entry until the date of the first new grade 3 or 4 adverse event. Participants lost to follow-up prior to reaching an adverse event endpoint or not documented to have reached an adverse event endpoint at the end of the study had their endpoint censored at the date of their last visit.
Time Frame: From study entry to week 72
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: cumulative probability per 100 persons
Arm/Group | CAP-IT | Standard Care
Number analyzed (Participants) | 86 | 86
cumulative probability per 100 persons | 6 [3 to 14] | 2 [1 to 9]

ADVERSE EVENTS:
Time Frame: From treatment dispensation until off-study at any time throughout the study (up to 213 weeks), participant follow-up time was variable
Description: There were no drugs administered through the study and SAEs were reported to local IRB/ECs only. The protocol requested recording of new signs and symptoms >=Grade 3, any AEs that led to a change in ART, regardless of grade, and all diagnoses identified according to ACTG criteria. DAIDS AE Grading Table (V1, 2004; Clarification 2009) was used.
Arm/Group | CAP-IT | Standard Care
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/86
Other Adverse Events (participants affected / at risk) | 44/86 | 38/86
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CAP-IT (N=86) | Standard Care (N=86)
Anaemia (Blood and lymphatic system disorders) | 9 | 6
Diarrhoea (Gastrointestinal disorders) | 8 | 4
Nausea (Gastrointestinal disorders) | 7 | 4
Hypertransaminasaemia (Hepatobiliary disorders) | 4 | 6
Drug hypersensitivity (Immune system disorders) | 30 | 23
Latent syphilis (Infections and infestations) | 5 | 3
Nasopharyngitis (Infections and infestations) | 7 | 5
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 8
Dizziness (Nervous system disorders) | 7 | 4
Headache (Nervous system disorders) | 7 | 3
Depression (Psychiatric disorders) | 9 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No